CLINICAL TRIAL: NCT01818128
Title: The Pretreatment of a Left-sided Double-lumen Tube to Prevent Its Misplacement to the Right Mainstem Bronchus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_DLT_flexion
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Double Lumen Tube Intubation

ARMS (2):
- Neutral shape of bronchial tip (Active Comparator)
  Interventions: Device: Neutral shape of bronchial tip
- Bent shape of bronchial tip (Experimental)
  Interventions: Device: Bent shape of bronchial tip

INTERVENTIONS:
Device: Neutral shape of bronchial tip — Intubation is performed without transforming the shape of the bonchial tipof a double lumen tube.
  Arms: Neutral shape of bronchial tip
Device: Bent shape of bronchial tip — Intubation is performed with the double lumen tube, which bronchial tip has been bent 45 degrees and maintained for 5 min.
  Arms: Bent shape of bronchial tip

SUMMARY:
The purpose of this study is to investigate whether flexion of bronchial tip of a left-sided double lumen endobronchial tube prevents tube misplacement to the right mainstem bronchus.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that require the placement of left-sided double-lumen tubes

Exclusion Criteria:

* Abnormal anatomy of tracheobronchial tree
* Intraluminal lesion in the left or right mainstem bronchus
* Anticipated difficult intubation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1540 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with intubation to right mainstem bronchus | An expected average of 5minutes after intubation

SECONDARY OUTCOMES:
Number of participants with airway injury | An expected average of 5 minutes after bilateral lung ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea